CLINICAL TRIAL: NCT04850027
Title: MAgnetic Resonance Imaging Guided LAteral Lymph Node Dissection in Lower REctal Cancer - A Multicenter, Prospective, Registry Study (MALAREC)
Brief Title: MRI-guided Lateral Lymph Node Dissection in Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Shengjing Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); China-Japan Friendship Hospital (Other); Peking University First Hospital (Other); Beijing Friendship Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University Cancer Hospital & Institute (Other); The First Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Tianjin People's Hospital (Other); Second Affiliated Hospital of Suzhou University (Other); Peking Union Medical College Hospital (Other); Ruijin Hospital (Other); First Hospital of China Medical University (Other); Chinese PLA General Hospital (Other); Zhejiang Cancer Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: MALAREC
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
Keywords: Lateral lymph node; Surgery; Magnetic resonance imaging; oncological outcome
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower rectal cancer patients with a LLN ≥ 5mm: Patients with lateral lymph node short diameter ≥ 5mm evaluated by MRI were included.
  Interventions: Procedure: TME+Lateral lymph node dissection.

INTERVENTIONS:
Procedure: TME+Lateral lymph node dissection. — TME and lateral lymph node dissection is performed in rectal cancer patients with lateral lymph node short diameter ≥ 5 mm.

SUMMARY:
To investigate the oncological outcome of lateral lymph node dissection in low rectal cancer based on MRI

DETAILED DESCRIPTION:
Our study design is a multicenter, prospective, registry study.

We would enroll 268 patients with lower rectal cancer whose preoperative MRI showed laterally lymph node diameter ≥ 5mm.

The postoperative adjuvant chemoradiotherapy is determined by the pathological results. For patients of stage II and patients of stage III with unfavorable histologic features, six months of adjuvant chemotherapy of fluorouracil-based regimen with radiotherapy of 45.0 ~ 50.5 Gy are recommended.

The postoperative examination should be performed every three months in the first two years and every six months in the following three years.

Our study is expected to last five years, of which two years for recruiting patients, three years for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old
2. Pathologically confirmed as rectal adenocarcinoma
3. The tumor is located in the middle or lower rectum
4. Preoperative MRI assessment is T2-4 N+M0
5. Lateral lymph node short diameter ≥ 5 mm (MRI)
6. Signed informed consent

Exclusion Criteria:

1. Previous history of malignant colorectal tumors
2. Multiple abdominal or pelvic surgeries were performed
3. Complicated with bowel obstruction, perforation or bleeding
4. Patients undergoing palliative surgery
5. Patients with severe liver and kidney dysfunction, cardiopulmonary dysfunction, blood coagulation dysfunction, or combined with serious underlying diseases that cannot tolerate surgery
6. Have a history of severe mental illness
7. Pregnant or breastfeeding women （8) Patients previously treated with iliac artery surgery (or its branches)

(9) R0 resection cannot complete (10) ASA grade ≥ IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower rectal cancer patients with lateral lymph node short diameter ≥ 5 mm were included in the study. TME with lateral lymph node dissection was performed in these patients. LLN positive rate, local recurrence rate, 3-year overall survival rate, perioperative complication rate and quality of life were documented and analysed.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological positive rate | 3-year.
  The proportion of patients with positive lateral lymph node which was confirmed pathologically.
Local recurrence rate | 3-year
  The proportion of patients with local recurrence after 3 years of surgery
Overall survival rate | 3-year
  The proportion of patients survived after 3 years of surgery
Disease free survival | 3-year
  The proportion of patients with no disease recurrence and metastasis after 3 years of surgery.

SECONDARY OUTCOMES:
Early morbidity rate | 30 days
  The early morbidity rate is defined as the event observed during operation and within 30 days after surgery
Duration of the surgery | 1 day
  The duration of time between the start and the end of the surgery.
Postoperative complications | 30 days
  Complications occurring within 30 days after surgery, mainly urinary and sexual functions.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Liu, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data are available from Qian Liu upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data were available to all the researchers permanently after this study was done.
Access Criteria: All the data will be available to all the relevant researchers in the world upon request. Email: liuqianncc@126.com

REFERENCES:
- [Background] Baik SH, Kim NK, Lee YC, Kim H, Lee KY, Sohn SK, Cho CH. Prognostic significance of circumferential resection margin following total mesorectal excision and adjuvant chemoradiotherapy in patients with rectal cancer. Ann Surg Oncol. 2007 Feb;14(2):462-9. doi: 10.1245/s10434-006-9171-0. Epub 2006 Nov 10. PMID 17096053
- [Background] Akiyoshi T, Ueno M, Matsueda K, Konishi T, Fujimoto Y, Nagayama S, Fukunaga Y, Unno T, Kano A, Kuroyanagi H, Oya M, Yamaguchi T, Watanabe T, Muto T. Selective lateral pelvic lymph node dissection in patients with advanced low rectal cancer treated with preoperative chemoradiotherapy based on pretreatment imaging. Ann Surg Oncol. 2014 Jan;21(1):189-96. doi: 10.1245/s10434-013-3216-y. Epub 2013 Aug 21. PMID 23963871
- [Background] Fujita S, Mizusawa J, Kanemitsu Y, Ito M, Kinugasa Y, Komori K, Ohue M, Ota M, Akazai Y, Shiozawa M, Yamaguchi T, Bandou H, Katsumata K, Murata K, Akagi Y, Takiguchi N, Saida Y, Nakamura K, Fukuda H, Akasu T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Mesorectal Excision With or Without Lateral Lymph Node Dissection for Clinical Stage II/III Lower Rectal Cancer (JCOG0212): A Multicenter, Randomized Controlled, Noninferiority Trial. Ann Surg. 2017 Aug;266(2):201-207. doi: 10.1097/SLA.0000000000002212. PMID 28288057
- [Background] Ishihara S, Kawai K, Tanaka T, Kiyomatsu T, Hata K, Nozawa H, Morikawa T, Watanabe T. Oncological Outcomes of Lateral Pelvic Lymph Node Metastasis in Rectal Cancer Treated With Preoperative Chemoradiotherapy. Dis Colon Rectum. 2017 May;60(5):469-476. doi: 10.1097/DCR.0000000000000752. PMID 28383446
- [Background] Furuhata T, Okita K, Nishidate T, Ito T, Yamaguchi H, Ueki T, Akizuki E, Meguro M, Ogawa T, Kukita K, Kimura Y, Mizuguchi T, Hirata K. Clinical feasibility of laparoscopic lateral pelvic lymph node dissection following total mesorectal excision for advanced rectal cancer. Surg Today. 2015 Mar;45(3):310-4. doi: 10.1007/s00595-014-0906-4. Epub 2014 May 3. PMID 24792010
- [Derived] Huang F, Wei R, Zhou S, Mei S, Xiao T, Xing W, Liu Q; the Chinese Lateral Node Collaborative Group. The diagnosis and oncological outcomes of obturator and internal iliac lymph node metastasis in middle-low rectal cancer: results of a multicenter Lateral Node Collaborative Group study in China. Discov Oncol. 2024 Nov 4;15(1):618. doi: 10.1007/s12672-024-01500-4. PMID 39497010
- [Derived] Tang B, Zhou S, He K, Mei S, Qiu W, Guan X, Liu F, Chi C, Wang X, Tian J, Liu Q, Tang J. Applications of Near-Infrared Fluorescence Imaging and Angiography of Inferior Vesical Artery in Laparoscopic Lateral Lymph Node Dissection: A Prospective Nonrandomized Controlled Study. Dis Colon Rectum. 2024 Jan 1;67(1):175-184. doi: 10.1097/DCR.0000000000002926. Epub 2023 Aug 30. PMID 38091416
- [Derived] Zhou S, Zhang H, Liang J, Fu W, Lou Z, Feng B, Yang Y, Xie Z, Liu Q; Chinese Lateral Node Collaborative Group. Feasibility, Indications, and Prognostic Significance of Selective Lateral Pelvic Lymph Node Dissection After Preoperative Chemoradiotherapy in Middle/Low Rectal Cancer: Results of a Multicenter Lateral Node Study in China. Dis Colon Rectum. 2024 Feb 1;67(2):228-239. doi: 10.1097/DCR.0000000000002640. Epub 2023 Jan 4. PMID 36649192
- [Derived] Zhou S, Mei S, Feng B, Yang Y, Wang X, Wang Q, Liu Q. Feasibility and safety of lateral pelvic lymph node dissection for elderly patients with middle-low rectal cancer: results of a large multicenter lateral node collaborative group study in China. Tech Coloproctol. 2023 Aug;27(8):655-664. doi: 10.1007/s10151-022-02746-2. Epub 2022 Dec 14. PMID 36515808
- [Derived] Zhou S, Tang J, Liang J, Lou Z, Fu W, Feng B, Yang Y, Xiao Y, Liu Q. Effective dissecting range and prognostic significance of lateral pelvic lymph node dissection for middle-low rectal cancer patients with lateral pelvic lymph node metastasis: Results of a large multicenter lateral node collaborative group in China. Front Oncol. 2022 Aug 12;12:916285. doi: 10.3389/fonc.2022.916285. eCollection 2022. PMID 36033473
- [Derived] Zhou S, Song Y, Xie Y, Liu Q. Neoadjuvant Chemoradiotherapy Prior to Lateral Lymph Node Dissection in Rectal Cancer with Suspected Lateral Lymph Node Metastasis: a Multicenter Lateral Node Study in China. J Gastrointest Surg. 2023 Jan;27(1):158-161. doi: 10.1007/s11605-022-05425-7. Epub 2022 Jul 26. No abstract available. PMID 35882759